CLINICAL TRIAL: NCT00459212
Title: Phase I and Pharmacodynamic Study of GTI-2040 (NSC 722929, IND 67368) in Acute Leukemias
Brief Title: GTI-2040 in Treating Patients With Relapsed, Refractory, or High-Risk Acute Leukemia, High-Grade Myelodysplastic Syndromes, or Refractory or Blastic Phase Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00206; PHI-57; CDR0000539257; U01CA062505 (NIH)
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2013-04

CONDITIONS: Acute Undifferentiated Leukemia; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Blastic Phase Chronic Myelogenous Leukemia; de Novo Myelodysplastic Syndromes; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Untreated Adult Acute Lymphoblastic Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Congenital Abnormalities; Blast Crisis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — GTI2040

ARMS (1):
- Arm I (Experimental): Patients receive GTI-2040 IV continuously on days 1-4 and 15-18.
  Interventions: Drug: GTI-2040; Procedure: pharmacological study; Procedure: laboratory biomarker analysis

INTERVENTIONS:
Drug: GTI-2040 — Given IV
Procedure: pharmacological study — Correlative study
  Other Names: pharmacological studies
Procedure: laboratory biomarker analysis — Correlative study

SUMMARY:
This phase I trial is studying the side effects and best dose of GTI-2040 in treating patients with relapsed, refractory, or high-risk acute leukemia, high-grade myelodysplastic syndromes, or refractory or blastic phase chronic myelogenous leukemia. Drugs used in chemotherapy, such as GTI-2040, work in different ways to stop the growth of cancer or abnormal cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of GTI-2040 in patients with relapsed, refractory, or high-risk acute leukemia, high-grade myelodysplastic syndromes, or refractory or blastic phase chronic myelogenous leukemia.

II. Assess the toxicity and efficacy of this drug in these patients. III. Assess plasma and intracellular pharmacokinetics of this drug in these patients.

OUTLINE: This is a multicenter, dose-escalation study.

Patients receive GTI-2040 IV continuously on days 1-4 and 15-18. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of GTI-2040 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Blood samples are collected on days 1, 4, 15, and 19 of course 1 for pharmacokinetic studies. Samples are analyzed by proteomic assay, dCTP pool measurement, and real-time polymerase chain reaction for mRNA of RRM2, RRM1, and p53R2.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 1 of the following:

  * Acute myeloid leukemia (AML) or acute lymphoblastic leukemia (ALL) refractory to primary standard induction therapy
  * Relapsed or refractory acute leukemia
  * Chronic myelogenous leukemia (CML) in blast crisis at diagnosis OR that failed prior aggressive induction chemotherapy
* Diagnosis of 1 of the following:

  * Acute leukemia secondary to preexisting hematologic condition or prior chemotherapy at diagnosis OR that failed prior aggressive induction chemotherapy
  * Advanced myelodysplastic syndromes (intermediate-1 or greater)
  * De novo acute leukemia (myeloid or nonmyeloid)
* Not a candidate for aggressive standard induction chemotherapy
* De novo AML or ALL (patients > 60 years of age)
* No suspected or proven active CNS leukemia
* ECOG performance status (PS) 0-2 OR Karnofsky PS 50-100%
* Life expectancy >= 8 weeks
* Bilirubin =< 1.5 mg/dL
* AST and ALT < 3 times upper limit of normal (ULN)
* Creatinine =< 1.5 times ULN
* No HIV positivity
* Fertile patients must use effective contraception
* No history of allergic reactions attributed to other phosphorothiolated oligonucleotides
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing, active, or poorly controlled infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Cardiac arrhythmia
  * Poorly controlled pulmonary disease
  * Psychiatric illness or social situation that would preclude study compliance
* Recovered from all prior therapies
* Prior autologous or allogeneic stem cell transplantation allowed (No active graft-vs-host disease > grade 2)
* At least 2 weeks since prior and no concurrent cytotoxic chemotherapy
* At least 2 weeks since prior and no concurrent biologic therapy
* At least 2 weeks since any other prior investigational agent
* No other concurrent anticancer therapy, including radiotherapy or hormonal therapy
* Concurrent imatinib mesylate for CML allowed
* Not pregnant or nursing
* Negative pregancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-03; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) determined according to dose-limiting toxicities (DLTs) graded using Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0) | 28 days
Change in dCTP levels in PBMC and bone marrow by Real-Time PCR | Days 1, 4, 15, and 19 of course 1

SECONDARY OUTCOMES:
Objective tumor response | Up to 3 years
Overall survival | Up to 3 years
Time to failure | Up to 3 years
Duration of response | Up to 3 years
Change in expression levels of R1, R2, and p53R2 mRNA in PBMC by Real-Time PCR | Day 1, 4, 15, and 19 of course 1
Change in intracellular levels of GTI-2040 by ELISA | Day 1, 4, 15, and 19 of course 1
Incidence of grade 3 or higher toxicity assessed by CTCAE v3.0 | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kirschbaum, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States